CLINICAL TRIAL: NCT03673865
Title: Does the Use of a Customized Titanium Reconstruction Plate for Orbital Fractures Result in Better Orbital Volume and Outcome
Brief Title: The Use of 3D Printing in Orbital Fractures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment and study activities were initially suspended due to COVID-19 and it has been determined that the study will not resume.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Dina Amin, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00103655
Record Dates: First submitted 2018-09-14; First posted 2018-09-17 (Actual); Results first posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Orbital Fractures
Keywords: 3D Printer; orbital implants
MeSH Terms: conditions — Orbital Fractures

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized clinical study with longitudinal follow-up
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment Group (Experimental): Patients undergo orbital reconstruction using pre-adjusted patient-specific orbital implants with office-based 3-dimensional printers (OB3DP)
  Interventions: Device: office-based 3-dimensional printers (OB3DP)
- Control Group (Active Comparator): Patients undergo orbital reconstruction with non-patient-specific orbital implants (traditional approach, Control Group) which is a standard stock orbital plate
  Interventions: Device: standard stock orbital plate

INTERVENTIONS:
Device: office-based 3-dimensional printers (OB3DP) — In this treatment group subjects, using office-based 3-dimensional printers (OB3DP) a patient-specific pre-adjusted (pre-bend) orbital plates will be made using over-the-counter titanium plates that are manually adjusted according to the printed model. The plates are then send to sterilization for preparation.
  Other Names: 3D Printer; Prusa i3 MK2 3D Printer kit with liquid crystal display
  Arms: Treatment Group
Device: standard stock orbital plate — In this control group subjects will receive non-patient-specific orbital implants which is standard stock orbital plate that is adapted intraoperatively to the fractured orbit
  Other Names: orbital plate
  Arms: Control Group

SUMMARY:
The study is a prospective randomized longitudinal clinical study to compare pre-adapted patient-specific orbital implants utilizing an office-based 3-D printer versus standard non-adapted orbital implants (the latter being the traditional approach and current standard of care).

DETAILED DESCRIPTION:
Orbital fracture, which accounts for 10-25% of facial fractures, is one of the most difficult facial fractures to treat. The complex bone anatomy and the proximity of adjacent vital structures make reconstruction of these fractures challenging. Inadequate orbital fracture reconstruction leads to cosmetic and functional complications. Cosmetic complications include enophthalmos, which is defined as posterior displacement of the eyeball within the orbit due to changes in the volume of the orbit (bone) relative to its contents (the eyeball and orbital fat). Functional complications include diplopia, defined as a type of vision disorder in which two images are seen of a single object.

This is a prospective randomized clinical study with longitudinal follow-up. The study duration is 2 years, and it will be conducted at Grady Memorial Hospital (GMH). The study targets low-income, urban adults suffering blunt facial trauma who are diagnosed with unilateral orbital fracture.

The purpose of this study is to compare pre-adapted patient-specific orbital implants utilizing an office-based 3-D printer versus standard non-adapted orbital implants. Main aims of the study are to 1) preoperatively generate a patient-specific model to pre-adapt the titanium mesh for use in unilateral orbital fractures; 2) accurately restore the orbital volume to pre-injury levels; 3) prevent postoperative complications including enophthalmos and diplopia; and 4) decrease the operative time, therefore decreasing overall cost and increasing value.

ELIGIBILITY:
Inclusion Criteria:

* Agreed to be enrolled in the study.
* Indications for surgical repair of orbital floor and/ wall fractures are dependent on several factors:

  * Correction or prevention of cosmetic deformity ( enophthalmos or inferior dystopia; disruption of greater than 50% of the orbital floor is likely to cause cosmetically apparent enophthalmos.
  * Correction of unresolved diplopia (7 to 11 days) in the sitting of soft tissue prolapse with a positive forced duction test.
  * Immediate correction of diplopia in the sitting inferior rectus muscle incarceration and a positive forced duction test.
  * Immediate correction in a symptomatic patient with orbital floor ( trapdoor) fracture that has elicited the oculocardiac reflex.
* At least 18 years of age.
* Unilateral orbital floor fracture.
* No history of orbital trauma.
* Healthy contralateral orbit.
* Underwent orbital reconstruction.
* Admitted to GMH.
* Returned for the 6-week follow-up.

Exclusion Criteria:

* Refuse study enrollment.
* Are younger than 18 years.
* Pregnant women.
* Prisoner
* Unable to obtain consent (cognitively impaired)
* Are admitted to hospitals other than Grady Memorial Hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dina Amin, DDS, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group | Control Group
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Control Group | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 41.5 [21 to 63] | 38.2 [18 to 69] | 39.9 [23 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 7 | 8 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 3 | 1 | 4
  Other | 1 | 0 | 1
  African-American | 9 | 11 | 20
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 25
Medical Comorbidities [Count of Participants; unit: Participants]
  Hypertension | 6 | 4 | 10
  Diabetes | 2 | 1 | 3
  Migraines | 2 | 0 | 2
  Asthma | 2 | 0 | 2
  Depression | 1 | 1 | 2
Etiology [Count of Participants; unit: Participants]
  MVC | 1 | 4 | 5
  Fall | 3 | 1 | 4
  Assault | 8 | 3 | 11
  Other | 1 | 4 | 5
Laterality [Count of Participants; unit: Participants]
  Left | 6 | 8 | 14
  Right | 7 | 4 | 11
Location of fracture [Count of Participants; unit: Participants]
  Orbital floor fracture | 11 | 12 | 23
  Medial wall fracture | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Orbital Volume of the Injured Orbit Compared to the Contralateral Uninjured Orbit as Assessed by CT Scan Between the Treatment and Control Groups
Description: The Primary Investigator will evaluate the orbital volume using OsiriX (medical software). Orbital volume measurements will be obtained to compare the injured and uninjured (contralateral) orbital volumes. OsiriX MD offers advanced processing techniques and has the ability to precisely measure orbital volume. It also utilizes the DICOM data from the immediate postoperative CT scans.
Time Frame: 1 hour post operatively
Measure: Mean (Standard Deviation); unit: Cm^3
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 13 | 12
Cm^3
  Uninjured Orbit | 23 (3.5) | 22.8 (2.6)
  Reconstructed Orbit | 23.5 (3.2) | 28.6 (3.6)

2. Secondary Outcome: Number of Subjects With Reduction of Orbital Volume to Less Than 2 cm3 Between the Treatment and Control Groups
Description: Adequate orbital volume reduction, defined as a reduction of orbital volume to less than 2 cm3. The Primary Investigator will evaluate the orbital volume using OsiriX (medical software). Number of subjects with reduction of orbital volume to less than 2 cm3 between the treatment and control groups are recorded
Time Frame: 1 week, 3 weeks, and 6 weeks postoperatively.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 13 | 12
Participants
  1 week postoperatively. | 13 | 12
  3 weeks postoperatively. | 13 | 12
  6 weeks postoperatively | 13 | 12

3. Secondary Outcome: Number of Subjects With a Difference of More Than 2 mm Between the Two Orbits Between the Treatment and Control Groups
Description: A difference of more than 2 mm between the two orbits is diagnostic for enophthalmos. Enophthalmos is assessed by clinical examination using a Hertel exophthalmometer. The measurement is taken from the lateral orbital rim to the corneal apex. The normal range is 12-21 mm. Upper normal limit for people of African origin is a little higher, about 23-24 mm. A difference greater than 2 mm between the eyes is significant.
Time Frame: 1 week, 3 weeks, and 6 weeks postoperatively.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 13 | 12
Participants
  1 week postoperatively. | 0 | 0
  3 weeks postoperatively. | 0 | 0
  6 weeks postoperatively. | 0 | 0

4. Secondary Outcome: Number of Subjects With Infection Between the Treatment and Control Groups
Description: Infection is defined by the presence of postoperative pus in the wound, a sinus tract or fistula, or elevated white blood cell count (WBC) >11.0x109/L combined with erythematous skin and swelling on the operated side more than on the un-operated side. WBC is measured with a blood draw test. Infection will be confirmed with clinical examination along with blood tests.
Time Frame: 1 week, 3 weeks, and 6 weeks postoperatively.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 13 | 12
Participants
  1 week postoperatively. | 0 | 0
  3 weeks postoperatively. | 0 | 0
  6 weeks postoperatively. | 0 | 0

5. Secondary Outcome: Number of Subjects With Infraorbital Nerve Injury Between the Treatment and Control Groups
Description: Infraorbital nerve injury is assessed by clinical examination using neurosensory testing (NST). NST is a standardized methodology designed to objectively evaluate sensory nerve function. The sensory impairment is determined by 3 levels of testing; each level classifies a specific type of sensory nerve injury.
Time Frame: 1 week, 3 weeks, and 6 weeks postoperatively.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 13 | 12
Participants
  1 week postoperatively. | 0 | 0
  3 weeks postoperatively. | 0 | 0
  6 weeks postoperatively. | 0 | 0

6. Secondary Outcome: Number of Subjects With Intraocular Pressure (IOP) > 40 mmHg Between the Treatment and Control Groups
Description: Intraocular pressure (IOP) > 40 mmHg is diagnostic of orbital compartment syndrome. Orbital compartment syndrome is assessed through clinical examination using tonometry test. Tonometry is a diagnostic test that measures the pressure inside your eye, which is called intraocular pressure (IOP). The normal pressure range is 12 to 22 mm Hg.
Time Frame: 1 week, 3 weeks, and 6 weeks postoperatively.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 13 | 12
Participants
  1 week postoperatively. | 0 | 0
  3 weeks postoperatively. | 0 | 0
  6 weeks postoperatively. | 0 | 0

7. Secondary Outcome: Mean Operating Time in Minutes Between the Treatment and Control Groups
Description: Operating time will be calculated from fracture exposure and identification to the final implant placement and fixation and will be recorded in minutes. This will be compared between the two treatment groups. To record and compare the operative time between the two groups, a stopwatch will be utilized.
Time Frame: Intraoperative time period
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 13 | 12
minutes
  Length of surgery | 32.6 (13.7) | 53.3 (12.8)
  Time interval from plate insertion to fixation | 15.8 (14.4) | 41.4 (9.4)

8. Secondary Outcome: Mean Length of Stay in Hospital Measured in Days Between the Treatment and Control Groups
Description: Isolated orbital floor fracture patients do not require a pre-operative hospital stay. Length of stay will be calculated in terms of postoperative hospital stay (days). Length of stay in cases of complex orbital fracture will be calculated in terms of pre-operative and postoperative hospital stay (days). The number of days subject stays in the hospital are measured and compared
Time Frame: up to 2 weeks
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 13 | 12
days | 1.4 [0 to 5] | 2.1 [0 to 7]

9. Secondary Outcome: Mean Treatment Amount in Dollars Between the Treatment and Control Groups
Description: Treatment charges will be calculated with consideration of the following:
  1. Facility operating room charges, which include anesthesia time (surgical time multiplied by the facility rate of $33/ minute).
  2. Hardware charges (plates and screws).
  3. Length Of Stay charges (LOS multiplied by the facility daily rate of $1,690/ day).
  4. The cost of the 3D printed model including the cost of the 3D printer and filaments ($1.5).
  All treatment charge variables will be provided by the Grady Memorial Hospital Financial Planning and Analysis center. Total treatment charges facility operating room charges, hardware charges, LOS, and the 3D printed model cost will be compared between groups in a manner similar to that outlined in previous studies by our group.
Time Frame: up to 2 weeks
Measure: Mean (Standard Deviation); unit: US Dollars
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 13 | 12
US Dollars
  Cost of Operation Room | 992.54 (524.63) | 1,757.25 (422.64)
  3D Cost | 80 (0) | 0 (0)
  Length of Stay, Cost | 1690 (0) | 1690 (0)
  Cost of plate and screws | 840 (0) | 840 (0)
  Total Cost | 3602.54 (524.63) | 4287.25 (422.64)

10. Secondary Outcome: Number of Subjects That Develop Restricted Extraocular Motility That Was Not Present Before Between the Treatment and Control Groups
Description: Extra-ocular motility is assessed through clinical examination. The patient should be able to move the eyes through the six cardinal positions of gaze (left, right, up and right, up and left, down and right, down and left). All patients will be examined for the following:
  1. Development of restricted extraocular motility that was not present prior to the surgery.
  2. Persistent restriction of extraocular motility after the surgery
Time Frame: 1 week, 3 weeks, and 6 weeks postoperatively.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 13 | 12
Participants
  1 week postoperatively. | 0 | 0
  3 weeks postoperatively. | 0 | 0
  6 weeks postoperatively. | 0 | 0

11. Secondary Outcome: Number of Subjects With Inability to Achieve the Normal Orbital Contour Between the Treatment and Control Groups
Description: Inability to achieve the normal orbital contour as assessed in the immediate post-operative Computerized Tomography (CT) scan. Maxillofacial non-contrast CT scans according to the protocol will be obtained as part of the standard of care in managing orbital fractures and will be obtained for all subjects post operatively.
Time Frame: Up to 6 hours postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 13 | 12
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 6 weeks post-operatively
Arm/Group | Treatment Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 0/13 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-04): https://cdn.clinicaltrials.gov/large-docs/65/NCT03673865/Prot_SAP_001.pdf